CLINICAL TRIAL: NCT03647202
Title: An Open-label, Randomized, 3-period, 3-treatment Crossover Study to Evaluate the Effect of High-fat, High-calorie Food and Standard Food on the Single-dose Pharmacokinetics of Milademetan in Healthy Subjects
Brief Title: Food Effects on Milademetan Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DS3032-A-U115
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-09

CONDITIONS: Food Effects on Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to 1 of 6 treatment sequences (Sequences ABC, ACB, BAC, BCA, CAB, or CBA), according to a pre-generated randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence ABC (Experimental): Participants receive milademetan in a fasted condition (A), then with a high-calorie, high-fat breakfast (B), then with a standard breakfast (C) - with a washout period between treatments.
  Interventions: Drug: Milademetan Treatment A; Drug: Milademetan Treatment B; Drug: Milademetan Treatment C
- Sequence ACB (Experimental): Participants receive milademetan in a fasted condition (A), then with a standard breakfast (C), then with a high-calorie, high-fat breakfast (B) - with a washout period between treatments.
  Interventions: Drug: Milademetan Treatment A; Drug: Milademetan Treatment B; Drug: Milademetan Treatment C
- Sequence BAC (Experimental): Participants receive milademetan with a high-calorie, high-fat breakfast (B), then in a fasted condition (A), then with a standard breakfast (C) - with a washout period between treatments.
  Interventions: Drug: Milademetan Treatment A; Drug: Milademetan Treatment B; Drug: Milademetan Treatment C
- Sequence BCA (Experimental): Participants receive milademetan with a high-calorie, high-fat breakfast (B), then with a standard breakfast (C), then in a fasted condition (A) - with a washout period between treatments.
  Interventions: Drug: Milademetan Treatment A; Drug: Milademetan Treatment B; Drug: Milademetan Treatment C
- Sequence CAB (Experimental): Participants receive milademetan with a standard breakfast (C), then in a fasted condition (A), then with a high-calorie, high-fat breakfast (B) - with a washout period between treatments.
  Interventions: Drug: Milademetan Treatment A; Drug: Milademetan Treatment B; Drug: Milademetan Treatment C
- Sequence CBA (Experimental): Participants receive milademetan with a standard breakfast (C), then with a high-calorie, high-fat breakfast (B), then in a fasted condition (A) - with a washout period between treatments.
  Interventions: Drug: Milademetan Treatment A; Drug: Milademetan Treatment B; Drug: Milademetan Treatment C

INTERVENTIONS:
Drug: Milademetan Treatment A — Treatment A: Single oral dose of milademetan 160 mg capsules under fasted conditions
  Other Names: Experimental product
Drug: Milademetan Treatment B — Treatment B: Single oral dose of milademetan 160 mg capsules with a high-calorie, high-fat meal
  Other Names: Experimental product
Drug: Milademetan Treatment C — Treatment C: Single oral dose of milademetan 160 mg capsules with a standard meal.

SUMMARY:
The primary objectives of this trial are:

* To evaluate the effect of a high-calorie, high-fat meal on the single-dose pharmacokinetics (PK) of milademetan
* To evaluate the effect of a standard meal on the single-dose PK of milademetan

The key secondary objective is to evaluate the safety and tolerability of single-dose milademetan in all treatments.

The duration of the study for each individual participant will be approximately 8 weeks from the start of Screening (within 28 days prior to dosing of study drug on Day 1) through the final Follow-up visit or phone call. Participants will remain in the Clinical Research Unit (CRU) from Study Day -2 through Study Day 20 (a total of 22 days and 21 nights).

Participants will receive 3 single doses of study drug (at least 1 week apart) over the course of 15 days.

At the investigator's discretion, participants may be asked to return to the CRU 14 days (±2 days) after final dose of study drug for a follow-up visit.

The end of the study is defined as the date of final follow-up visit of the last subject undergoing the study.

ELIGIBILITY:
Healthy participants with no clinically significant medical history or physical examination findings and who also meet all protocol-defined inclusion and exclusion criteria summarized as follows:

Inclusion Criteria:

* Has negative urine test for drugs of abuse, alcohol and tobacco
* If female, is surgically sterile or postmenopausal
* If male, agrees to protocol-defined contraceptive methods
* Has adequate hematologic, hepatic, and renal function as defined by the protocol
* Is able and willing to follow all study procedures
* Has provided a signed informed consent

Exclusion Criteria:

* Is female who is pregnant or breastfeeding
* Is unable to swallow oral medication
* Is unable to follow study procedures
* Has creatinine clearance < 90 mL/min at screening
* Is taking or has taken any medications or therapies outside of protocol-defined parameters
* Has history of or a known allergic reaction to azole antifungal agents
* Has any disease or condition that, per protocol or in the opinion of the investigator, might affect:

  1. safety and well-being of the participant or offspring
  2. safety of study staff

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of milademetan | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours postdose in each treatment period
Area under the plasma concentration-time curve (AUC) extrapolated to infinity (AUCinf) for milademetan | within 120 hours postdose in each treatment period

SECONDARY OUTCOMES:
Time to teach maximum plasma concentration (Tmax) of milademetan | within 120 hours postdose in each treatment period
AUC from time 0 to the time of last measurable concentration (AUClast) for milademetan | within 120 hours postdose in each treatment period
Lag time (tlag) for milademetan | within 120 hours postdose in each treatment period
  Tlag is used to characterize the delay in absorption of orally administered drugs
Terminal elimination half-life (t½) of milademetan | within 120 hours postdose in each treatment period
Apparent total body clearance (CL/F) of milademetan clearance (CL/F), | within 120 hours postdose in each treatment period
Apparent volume of distribution (Vz/F) of milademetan | within 120 hours postdose in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Covance Clinical Research Unit, Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/